CLINICAL TRIAL: NCT02107053
Title: The Effect of Pomegranate Juice on Oxidative Stress Biomarkers During Treatment With IV Iron During One Dialysis Session
Brief Title: The Effect of Pomegranate Juice (PJ) on Oxidative Stress Biomarkers During Treatment With IV Iron During One Dialysis Session
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Western Galilee Hospital-Nahariya (Other Government)
Collaborators: Luoxis (Industry)
Responsible Party: Principal Investigator, shifra sela, Head of Research Labs, Western Galilee Hospital-Nahariya
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 0122-13
Record Dates: First submitted 2014-02-18; First posted 2014-04-08 (Estimated); Last update posted 2016-02-09 (Estimated); Status verified 2016-02

CONDITIONS: Cardiovascular Disease (CVD)
Keywords: Oxidative stress,; hemodialysis,; pomegranate juice,; dietary supplement; patients
MeSH Terms: conditions — Cardiovascular Diseases | interventions — ferryl iron

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- IV iron + PJ (Experimental): Each patient will serve as a self control
  Interventions: Dietary Supplement: PJ; Drug: IV iron
- No IV iron + PJ (Experimental): Each patient will serve as a self control
  Interventions: Dietary Supplement: PJ
- IV iron no PJ (Experimental): Each patient will serve as a self control
  Interventions: Drug: IV iron

INTERVENTIONS:
Dietary Supplement: PJ
  Other Names: pomegranate juice
  Arms: IV iron + PJ; No IV iron + PJ
Drug: IV iron — IV iron is routinely administered to dialysis patients worldwide to correct anemia
  Arms: IV iron + PJ; IV iron no PJ

SUMMARY:
Atherosclerosis and its related cardiovascular morbidity and mortality, underlie many chronic diseases. Most atherosclerotic patients have multiple cardiovascular risk factors, which potentiate each other, causing a huge burden on health systems. In order to improve the understanding and treatment options of atherosclerosis, it is necessary to identify common basic pathways in its pathogenesis. Oxidative Stress (OS) has a major role in the pathogenesis of atherosclerosis; however, good biomarkers to determine OS are still missing.

DETAILED DESCRIPTION:
Cardiovascular disease (CVD) is a major cause of mortality and morbidity in industrialized countries. CVD associated with atherosclerosis is the major cause of death in patients treated with hemodialysis (HD) in addition to the high morbidity and mortality due to infections. Beside the invaluable goal of improving patients' quality of life, the reduction of the high prevalence of CVD leads to a significant financial consequences by lowering the financial burden on health systems.

Recently, the investigators have reported that half a cup of pomegranate juice (PJ), exceptional for its highest levels of antioxidants, administered 3 times a week for one year at the beginning of each dialysis, had many beneficial effects. The PJ led to a significant reduction of the atherosclerotic process and the rate of hospitalization due to infections: It lowered traditional CV risk factors such as high blood pressure and lipids (triglycerides levels). It improved various systemic non-traditional cardiovascular risk factors such as neutrophil priming, oxidation adducts and pro-inflammatory factors (IL-6, TNFα). Neutrophil priming was previously reported by us as a unique non-traditional CV risk factor involved in different clinical states associated with atherosclerosis. Moreover, the investigators have shown that primed neutrophils separated from HD patients cause endothelial injury that may lead to atherosclerosis and CVD.

The PJ is, thus, effective, vital and important. Yet the PJ in its natural liquid state has an astringent taste and raises doubts and uncertainties with regards to its non-standardized commercial preparation, of undefined composition and shelf life.

The investigators propose to examine PJ or pomegranate extracts containing similar concentrations of total polyphenols as in the investigators previous study in the Turkish juice (ref #2 below), in order to make it more standardized as a dietary supplement to hemodialysis patients.

The investigators plan in this protocol to study the effects of a chosen pomegranate extracts or juice from Primor, in a clinical study in HD patients. The study will be performed in one dialysis session, with and without IV iron and with and without pomegranate juice (4-arms, same patient). Each dialysis session activates neutrophils and induces oxidative stress and inflammation. Therefore, in this clinical study the investigators will assay the beneficial effects of the PJ on oxidative stress and inflammation induced by one dialysis session exacerbated by IV iron.

Each patient will be treated the same day of the week, 4 times, altogether one month per patient.

ELIGIBILITY:
Inclusion Criteria:

* patients on hemodialysis

Exclusion Criteria:

* patients with infections or cancer

Ages: 20 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2014-04; Primary Completion 2015-10 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Oxidation reduction potential | Immediately before and after dialysis, for 4 various protocols
  Each patient will serve as a self control. The metric measurements will be expressed as relative to control potential. Redox potential will be measured as oxidation-reduction potential and reported in millivolts.

CONTACTS AND LOCATIONS:
Overall Officials: Batya Kristal, MD, Principal Investigator — Western Galilee Hospital
Locations (1):
- Western Galilee Hospital, Nahariya, Israel

REFERENCES:
- [Background] Shema-Didi L, Kristal B, Ore L, Shapiro G, Geron R, Sela S. Pomegranate juice intake attenuates the increase in oxidative stress induced by intravenous iron during hemodialysis. Nutr Res. 2013 Jun;33(6):442-6. doi: 10.1016/j.nutres.2013.04.004. Epub 2013 May 9. PMID 23746559
- [Background] Shema-Didi L, Sela S, Ore L, Shapiro G, Geron R, Moshe G, Kristal B. One year of pomegranate juice intake decreases oxidative stress, inflammation, and incidence of infections in hemodialysis patients: a randomized placebo-controlled trial. Free Radic Biol Med. 2012 Jul 15;53(2):297-304. doi: 10.1016/j.freeradbiomed.2012.05.013. Epub 2012 May 17. PMID 22609423
- [Background] Sela S, Michelis R, Kristal B. Are oxidative modifications of proteins a metabolomic signature of cardiovascular disease in CKD? Am J Kidney Dis. 2013 Feb;61(2):350-1. doi: 10.1053/j.ajkd.2012.10.022. No abstract available. PMID 23318016
- [Background] Cohen-Mazor M, Sela S, Mazor R, Ilan N, Vlodavsky I, Rops AL, van der Vlag J, Cohen HI, Kristal B. Are primed polymorphonuclear leukocytes contributors to the high heparanase levels in hemodialysis patients? Am J Physiol Heart Circ Physiol. 2008 Feb;294(2):H651-8. doi: 10.1152/ajpheart.00952.2007. Epub 2007 Nov 21. PMID 18032524
- [Background] Mazor R, Kristal B, Cohen-Mazor M, Yagil C, Yagil Y, Sela S. The polymorphonuclear leukocyte contributes to the development of hypertension in the Sabra rat. J Hypertens. 2007 Nov;25(11):2249-56. doi: 10.1097/HJH.0b013e3282dd79b6. PMID 17921819
- [Background] Mazor R, Shurtz-Swirski R, Farah R, Kristal B, Shapiro G, Dorlechter F, Cohen-Mazor M, Meilin E, Tamara S, Sela S. Primed polymorphonuclear leukocytes constitute a possible link between inflammation and oxidative stress in hyperlipidemic patients. Atherosclerosis. 2008 Apr;197(2):937-43. doi: 10.1016/j.atherosclerosis.2007.08.014. Epub 2007 Sep 17. PMID 17869258
- [Background] Jacobi J, Sela S, Cohen HI, Chezar J, Kristal B. Priming of polymorphonuclear leukocytes: a culprit in the initiation of endothelial cell injury. Am J Physiol Heart Circ Physiol. 2006 May;290(5):H2051-8. doi: 10.1152/ajpheart.01040.2005. Epub 2005 Dec 30. PMID 16387791
- [Background] Jacobi J, Kristal B, Chezar J, Shaul SM, Sela S. Exogenous superoxide mediates pro-oxidative, proinflammatory, and procoagulatory changes in primary endothelial cell cultures. Free Radic Biol Med. 2005 Nov 1;39(9):1238-48. doi: 10.1016/j.freeradbiomed.2005.06.010. Epub 2005 Aug 8. PMID 16214039
- [Background] Sela S, Shurtz-Swirski R, Cohen-Mazor M, Mazor R, Chezar J, Shapiro G, Hassan K, Shkolnik G, Geron R, Kristal B. Primed peripheral polymorphonuclear leukocyte: a culprit underlying chronic low-grade inflammation and systemic oxidative stress in chronic kidney disease. J Am Soc Nephrol. 2005 Aug;16(8):2431-8. doi: 10.1681/ASN.2004110929. Epub 2005 Jun 29. PMID 15987755
- [Background] Sela S, Mazor R, Amsalam M, Yagil C, Yagil Y, Kristal B. Primed polymorphonuclear leukocytes, oxidative stress, and inflammation antecede hypertension in the Sabra rat. Hypertension. 2004 Nov;44(5):764-9. doi: 10.1161/01.HYP.0000144480.10207.34. Epub 2004 Sep 27. PMID 15452031
- [Background] Shurtz-Swirski R, Sela S, Herskovits AT, Shasha SM, Shapiro G, Nasser L, Kristal B. Involvement of peripheral polymorphonuclear leukocytes in oxidative stress and inflammation in type 2 diabetic patients. Diabetes Care. 2001 Jan;24(1):104-10. doi: 10.2337/diacare.24.1.104. PMID 11194213
- [Background] Kristal B, Shurtz-Swirski R, Chezar J, Manaster J, Levy R, Shapiro G, Weissman I, Shasha SM, Sela S. Participation of peripheral polymorphonuclear leukocytes in the oxidative stress and inflammation in patients with essential hypertension. Am J Hypertens. 1998 Aug;11(8 Pt 1):921-8. doi: 10.1016/s0895-7061(98)00099-5. PMID 9715783